CLINICAL TRIAL: NCT01435395
Title: Phase I Trial of Temozolomide, Bevacizumab Plus Bortezomib for Patients With Recurrent Glioblastoma Multiforme
Brief Title: Trial of Temozolomide, Bevacizumab Plus Bortezomib for Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Schering-Plough (Industry); Genentech, Inc. (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey James Olson, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00014595; WCI1837-10 (Other: Other)
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Bevacizumab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapy (Experimental): Therapy with temozolomide, bevacizumab and bortezomib
  Interventions: Drug: Temozolomide, bevacizumab and bortezomib

INTERVENTIONS:
Drug: Temozolomide, bevacizumab and bortezomib — Escalating temozolomide with standard dose bevacizumab and bortezomib

SUMMARY:
This is a single-center (Emory University), open-label, single arm, phase I study to assess safety and toxicity of bortezomib in combination with bevacizumab and escalating doses of temozolomide for patients with recurrent glioblastoma multiforme. Patients requiring anti-epileptic medications will have to be at least 10 days off EIAEDs. Only non-EIAEDs are accepted.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. Patients must have histologically confirmed diagnosis of a recurrent/progressive WHO grade IV malignant gliomas (glioblastoma multiforme and gliosarcoma).
3. Patients must have measurable progressive or recurrent disease by MRI within 2 weeks of starting treatment.
4. No prior bortezomib is allowed.
5. An interval of at least 6 weeks between prior surgical resection, 4 weeks from the end of prior radiotherapy.
6. Patients must be at least 10 days off any enzyme inducing anti-epileptic drugs (EIAEDs) of the cytochrome P450 (CYP-450) such as phenytoin, carbamazepine, phenobarbital.
7. Karnofsky performance status score of 60 or more.
8. Patients must have recovered from toxicity of prior therapy.
9. Hematocrit > 29%, absolute neutrophil count (ANC) > 1,500 cells/microliter, platelets > 125,000 cells/microliter for 14 days prior to treatment initiation.
10. Serum creatinine < 1.5 mg/dl, serum glutamic-oxaloacetic transaminase (SGOT) and bilirubin < 1.5 times upper limit of normal.
11. Prothrombin time/international normalized ratio (PT INR) < 1.4.
12. An interval of at least 3 months from the completion of most recent radiation therapy. At least 4 weeks from a non-nitrosourea chemotherapy regimen and at least 6 weeks from a nitrosourea containing regimen.
13. For patients on corticosteroids, they must have been on a stable dose for 1 week prior to entry if clinically recommended.
14. May have up to three biological therapies.
15. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
16. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
17. Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

1. Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
2. Greater than three prior recurrences.
3. Enzyme-inducing anti-epileptic drugs (EIAEDs) of the CYP-450 such as phenytoin, carbamazepine, phenobarbital.
4. Patients receiving concurrent investigational drugs.
5. Evidence of central nervous system (CNS) hemorrhage on baseline MRI or CT scan (except for grade 1 hemorrhage that has been stable for at least 3 months).
6. History of stroke within six months.
7. Requires therapeutic anti-coagulation.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics and psychiatric illness/social situations that would limit compliance with study requirements, or disorders associated with significant immunocompromised state.
9. Patient has a calculated or measured creatinine clearance of < 20 mL/minute within 14 days prior to treatment initiation.
10. Patient has greater or equal to Grade 2 peripheral neuropathy within 14 days before enrollment.
11. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (Appendix), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
12. Patient has hypersensitivity to bortezomib, boron, or mannitol.
13. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
14. Patient has received other investigational drugs within 14 days of treatment initiation
15. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
16. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy. Patients with prior malignancies must be disease free for at least 5 years.
17. Serious, non-healing wound, active ulcer, or untreated bone fracture. Bone fractures must be healed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Determination of progressive disease, complete or partial responses | 6 weeks
  Complete or partial responses will be based upon major changes in tumor size on the Gd-MRI scan compared to the baseline scan. Determination of progressive disease is based upon comparison to the previous scan with the smallest measurements.

SECONDARY OUTCOMES:
Assess the time to progression | 6 months
  Six month progression-free survival and overall survival of patients completing one cycle of the investigational therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Olson, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia